CLINICAL TRIAL: NCT05693519
Title: GastroIntestinal Cancer in Children and Adolescents (GICCA): a SEER Population-based Study
Brief Title: GastroIntestinal Cancer in Children and Adolescents
Acronym: GICCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Paul G. Kemps, MD (Other)
Collaborators: Juliana Children's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Paul G. Kemps, MD, Researcher, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Other Study IDs: nWMO-D4-2022-031
Record Dates: First submitted 2022-12-22; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Cancer; Colorectal Cancer; Gastric Cancer; Hepatoblastoma; Hepatocellular Carcinoma; Burkitt Lymphoma; Neuroendocrine Tumors
Keywords: SEER; Gastrointestinal; Cancer; Malignant; Child; Pediatric; Adolescent
MeSH Terms: conditions — Gastrointestinal Neoplasms; Colorectal Neoplasms; Stomach Neoplasms; Hepatoblastoma; Carcinoma, Hepatocellular; Burkitt Lymphoma; Neuroendocrine Tumors; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Patients aged 0-17 years at primary gastrointestinal cancer diagnosis
- Young people aged 18-24 years: Patients aged 18-24 years at primary gastrointestinal cancer diagnosis

SUMMARY:
The goal of this observational population-based cohort study is to investigate the clinical characteristics and outcomes of children and adolescents with primary gastrointestinal malignancies registered in the publicly available Surveillance, Epidemiology, and End Results (SEER) 17 database during 2000-2019.

DETAILED DESCRIPTION:
The investigators aim to describe the patient and tumor characteristics, treatments, and outcomes of children and adolescents diagnosed with primary gastrointestinal malignancies, and to analyze these data for trends over time. In addition, the investigators want to explore independent prognostic factors for overall survival. Finally, the investigators want to describe subsequent primary malignancies diagnosed among patients from the study cohort, as well as to calculate their risk of developing a second primary cancer relative to the general population. Data on children (aged 0-17 years at diagnosis) and young people aged 18-24 years at diagnosis are analyzed separately. Special focus is laid on patients with primary carcinomas of the gastrointestinal tract; particularly colorectal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age at primary gastrointestinal cancer diagnosis <25 years
* Diagnosis of a primary gastrointestinal malignancy as an individual's first primary malignancy

Exclusion Criteria:

* None

Ages: 0 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients aged 0-24 years with a diagnosis of a primary gastrointestinal malignancy as their first primary malignancy in the SEER 17 database from 2000 until (and including) 2019.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-06-22 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2000-2019
  Defined as the time between the date of diagnosis and the date of death from any cause (event) or date of last follow-up.

SECONDARY OUTCOMES:
Standardized incidence of second primary malignancies | 2000-2019
  Standardized incidence of second primary malignancies in patients who survived (i) two or more months, or (ii) five or more years after initial gastrointestinal cancer diagnosis, relative to the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Paul G. Kemps, MD, Principal Investigator — Leiden University Medical Center
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden, South Holland
  - Juliana Children's Hospital, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Data are publicly available through SEER under the SEER Research Data Use Agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Supporting information is available on reasonable request.
Access Criteria: When applicable, confidential information will be shared after a Data Transfer Agreement (DTA) has been signed by both parties.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT05693519/Prot_SAP_000.pdf